CLINICAL TRIAL: NCT01520454
Title: Differential Effects of Oral and Intravenous Lipid Administration on Leptin Signaling
Brief Title: Effect of Increased Free Fatty Acids on Leptin Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009P000370
Record Dates: First submitted 2012-01-04; First posted 2012-01-30 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Leptin Resistance
Keywords: Leptin resistance; Free fatty acids; Lipotoxicity
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride; soybean oil, phospholipid emulsion; Water; CD36 Antigens; Soybean Oil; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): IV saline with heparin, oral water
  Interventions: Drug: Saline; Dietary Supplement: Water; Drug: Heparin
- High dose fat solution (Experimental): Intralipid at high dose, with heparin and PO water
  Interventions: Drug: Intralipid; Dietary Supplement: Water; Drug: Heparin
- Low dose fat solution (Experimental): Low dose IV Intralipid with heparin and PO water
  Interventions: Drug: Intralipid; Dietary Supplement: Water; Drug: Heparin
- Oral fat (Experimental): Oral fat load with IV saline
  Interventions: Drug: Saline; Dietary Supplement: Water; Dietary Supplement: oral fat

INTERVENTIONS:
Drug: Saline — IV saline at 0.83 mL/kg/hr for six hours
  Arms: Oral fat; Placebo
Drug: Intralipid — Intralipid in either low-dose or high dose (10% vs. 20%) at 0.83 mL/kr/hr for six hours
  Other Names: intravenous lipids
  Arms: High dose fat solution; Low dose fat solution
Dietary Supplement: Water — Water by mouth
Dietary Supplement: oral fat — Soybean oil by mouth at 1.25 g/kg x 2 doses
  Other Names: soybean oil
  Arms: Oral fat
Drug: Heparin — Heparin bolus of 1000 units followed by 800 u/hr, adjust per partial thromboplastin time (PTT), for 5.5 hours
  Other Names: anti coated
  Arms: High dose fat solution; Low dose fat solution; Placebo

SUMMARY:
Obese people have elevated levels of the hormone leptin. Despite this, they seem to be resistant to the effects of this hormone, which usually regulates appetite and energy expenditure. This is similar to what happens with insulin levels in the obese. Furthermore, the way lipid ingestion versus lipid infusion may impact novel molecules secreted by tissues commonly affected in insulin resistant states such as liver and muscle have not yet been studied.

The aim of the present study is to investigate the effect of oral vs. different doses of IV lipid administration on molecular parameters related to glucose and energy homeostasis using a randomized, placebo-controlled design.

Additionally, we will examine how increased free fatty acids (FFAs) my impact intracellular leptin signaling such as the STAT3 pathway.

DETAILED DESCRIPTION:
We propose to test our hypotheses by conducting a non-blinded, interventional study evaluating the effects of acute leptin administration on intracellular leptin signaling pathways after a 6 hour infusion period comparing an oral high fat meal, high fat lipid infusion, low fat lipid infusion, or placebo infusion (saline)iv lipid infusion, placebo (saline) and oral high fat meal. After a screening visit, study participation involves 1 meal pick-up visit, 1 overnight visit, and one 1 follow-up visit. Subjects will be randomized to one of 4 groups: an oral high fat meal, fat emulsion 20% infusion , fat emulsion 10% infusion, and a placebo (saline) infusion infusion and an oral high fat meal.

We plan to screen 100 male and postmenopausal female subjects, with BMI greater than 18 kg/m2, to consent 60 in order to have 32-48 evaluable subjects, 8-12 subjects per group, completing all parts of the study.

The primary study outcome to be evaluated will be the changes in serum concentrations of glucose, hormones influencing metabolism such as insulin, fat-cell-secreted proteins such as leptin, molecules involved in metabolism such as free fatty acids (FFAs), and markers of inflammation such as interleukin (IL)-2 and interferon (IFN)-gamma.

The secondary outcome will be to examine the impacts of increased FFAs on intracellular leptin signaling by phosphorylation of STAT3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65

Exclusion Criteria:

1. Subjects with a history of any illness, other than obesity, that may affect insulin sensitivity (anemia, infectious diseases, renal or hepatic failure, uncontrolled hypertension, cancer, lymphoma, chronic inflammatory conditions such as inflammatory bowel disease and rheumatoid arthritis, states of cortisol or growth hormone excess, alcoholism or drug abuse, and eating disorders).
2. History of diabetes mellitus.
3. Subjects taking any medications that are known to influence glucose metabolism such as glucocorticoids will also be excluded. We will screen for these conditions by means of a detailed history and review of systems and physical examination (see below).
4. Subjects taking any medications known to affect lipids such as statins will also be excluded. We will screen for these similar to above.
5. Cholesterol greater or equal to 250 mg/dL and/or triglyceride levels greater than 500 mg/dL at the time of screening, as determined by laboratory testing.
6. Subjects who have a known history of anaphylaxis or anaphylactoid-like reactions or who have a known hypersensitivity to anesthetic agents such as Lidocaine or Marcaine will be excluded from the study.
7. Hypersensitivity to fat emulsion or any component of the formulation; severe egg or legume (soybean) allergies; pathologic hyperlipidemia, lipoid nephrosis, acute pancreatitis associated with hyperlipemia.
8. Hypersensitivity to heparin or any component of the formulation
9. Severe thrombocytopenia, uncontrolled active bleeding, disseminated intravascular coagulation (DIC); suspected intracranial hemorrhage.
10. Subjects with a history of bleeding dyscrasia, poor wound healing or any medical condition precluding supine position will be excluded from the study.
11. Unable to follow study protocol or any condition that in the opinion of the investigator makes the subject unsuitable for the study.
12. Pregnancy
13. Prior history of gastrectomy, gastric bypass surgery, or other weight loss surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, DSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Perakakis N, Kokkinos A, Angelidi AM, Tsilingiris D, Gavrieli A, Yannakoulia M, Tentolouris N, Mantzoros CS. Circulating levels of five proglucagon-derived peptides in response to intravenous or oral glucose or lipids and to a mixed-meal in subjects with normal weight, overweight, and obesity. Clin Nutr. 2022 Sep;41(9):1969-1976. doi: 10.1016/j.clnu.2022.07.001. Epub 2022 Jul 19. PMID 35961260
- See also: Mantzoros Lab Home Page — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Fat Solution: Intralipid at high dose, with heparin and PO water
  Intralipid: Intralipid in either low-dose or high dose (10% vs. 20%) at 0.83 mL/kr/hr for six hours
  Water: Water by mouth
  Heparin: Heparin bolus of 1000 units followed by 800 u/hr, adjust per PTT, for 5.5 hours
- Low Dose Fat Solution: Low dose IV Intralipid with heparin and PO water
  Intralipid: Intralipid in either low-dose or high dose (10% vs. 20%) at 0.83 mL/kr/hr for six hours
  Water: Water by mouth
  Heparin: Heparin bolus of 1000 units followed by 800 u/hr, adjust per PTT, for 5.5 hours
Period: Overall Study
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Started | 9 | 6 | 5 | 6
Completed | 9 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: IV saline with heparin, oral water
  Saline: IV saline at 0.83 mL/kg/hr for six hours
  Water: Water by mouth
  Heparin: Heparin bolus of 1000 units followed by 800 u/hr, adjust per PTT, for 5.5 hours
- Total: Total of all reporting groups
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat | Total
Number analyzed (Participants) | 9 | 6 | 5 | 6 | 26
Age, Customized [Median (Inter-Quartile Range); unit: years] | 35.3 [25.0 to 47.6] | 29.1 [24.2 to 38.7] | 48.6 [44.4 to 54.9] | 27.6 [24.2 to 46.9] | 35.2 [29.5 to 47.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 3 | 7
  Male | 7 | 5 | 4 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Circulating Glucagon-like Peptide-1 (GLP-1) Levels
Description: The GLP-1 area under the curve (AUC) was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas under the curve are presented
Measure: Mean (Standard Deviation); unit: pM*min
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
pM*min | 7147 (3547) | 11725 (4799) | 11898 (9996) | 28060 (8414)

2. Primary Outcome: Change in Circulating Gastric Inhibitory Polypeptide (GIP) Levels
Description: The GIP AUC fwas calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas under the curve are presented
Measure: Mean (Standard Deviation); unit: pM*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
pM*min/ml | 12894 (8803) | 11830 (4516) | 19386 (16823) | 60559 (36610)

3. Primary Outcome: Change in Circulating Ghrelin Levels
Description: The Ghrelin AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas under the curve are presented
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
pg*min/ml | 172886 (89970) | 129451 (46926) | 207863 (111684) | 166195 (110140)

4. Primary Outcome: Change in Circulating Peptide Tyrosine Tyrosine (PYY) Levels
Description: The PYY AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas under the curve are presented
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
pg*min/ml | 90016 (25755) | 65131 (14914) | 82474 (21072) | 144702 (27466)

5. Secondary Outcome: Change in Circulating Glucose Levels
Description: The Glucose AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas Under the Curve are presented
Measure: Mean (Standard Deviation); unit: mg*min/dl
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
mg*min/dl | 30683 (1249) | 28735 (1269) | 32566 (1531) | 31364 (869)

6. Secondary Outcome: Change in Circulating Insulin Levels
Description: The Insulin AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas Under the Curve are presented
Measure: Mean (Standard Deviation); unit: mU*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
mU*min/ml | 1765 (1555) | 2072 (970) | 2103 (1645) | 3021 (1426)

7. Secondary Outcome: Change in Circulating Leptin Levels
Description: The Leptin AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas Under the Curve are presented
Measure: Mean (Standard Deviation); unit: ng*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
ng*min/ml | 2050 (2233) | 3639 (4470) | 5439 (4671) | 4973 (5313)

8. Secondary Outcome: Change in Circulating Adiponectin Levels
Description: The Adiponectin AUC was calculated from baseline to six hours
Time Frame: Baseline to 6 hours
Population: Areas Under the Curve are presented
Measure: Mean (Standard Deviation); unit: ng*min/ml
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 9 | 6 | 5 | 6
ng*min/ml | 1546442 (500930) | 2273306 (1068651) | 1778846 (857433) | 1970601 (961699)

9. Secondary Outcome: Phosphorylation of STAT3 Pathways Downstream of Leptin After Lipid Administration
Description: Intracellular signaling mechanisms downstream of leptin (particularly the STAT3 pathway) in response to lipid administration as represented by phosphorylation (pSTAT3).
Time Frame: Baseline to 6 hours
Population: The analysis unfortunately can not be performed due to technical reasons as STAT3 was not able to be measured in the samples/not enough volume was left to perform the appropriate tests after trouble-shooting.
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | High Dose Fat Solution | Low Dose Fat Solution | Oral Fat
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No